CLINICAL TRIAL: NCT02081820
Title: Observational Study on the Prognostic Relevance of Admission Glycated Hemoglobin (HbA1C) in Patients With Aneurysmal Subarachnoid Hemorrhage
Brief Title: Admission HbA1C in Aneurysmal Subarachnoid Hemorrhage
Status: Completed | Type: Observational
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, Neurochirurgische Klinik, Universitätsklinikum Düsseldorf, Neurochirurgische Klinik, Universitätsklinikum Düsseldorf, Heinrich-Heine University, Duesseldorf
Other Study IDs: UKD-NCH-2014-001
Record Dates: First submitted 2014-02-28; First posted 2014-03-07 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Hyperglycemia; Aneurysmal Subarachnoid Hemorrhage
Keywords: hyperglycemia; aneurysmal subarachnoid hemorrhage; glycated hemoglobin; outcome; DCI
MeSH Terms: conditions — Hyperglycemia; Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- aneurysmal subarachnoid hemorrhage: observational, no intervention

SUMMARY:
In patients suffering from aneurysmal subarachnoid hemorrhage (aSAH), hyperglycemia is considered an adverse prognostic factor. Glycated hemoglobin (or HbA1c) can be measured to estimate the average plasma glucose concentration over prolonged periods of time, thus determination of glycated hemoglobin at admission after aSAH serves as an approximation of blood glucose levels in the weeks preceding aneurysm rupture. In this patient registry admission HbA1c, clinical course and neurological outcome after 6 month are recorded, to determine whether elevated blood glucose levels prior to aneurysm rupture influence the clinical course and patient outcome after aSAH.

DETAILED DESCRIPTION:
In patients suffering from aneurysmal subarachnoid hemorrhage (aSAH), hyperglycemia is considered an adverse prognostic factor. Glycated hemoglobin (or HbA1c) can be measured to estimate the average plasma glucose concentration over prolonged periods of time, thus determination of glycated hemoglobin at admission after aSAH serves as an approximation of blood glucose levels in the weeks preceding aneurysm rupture.

In this patient registry admission HbA1c within 72 hours after confirmed aneurysmal subarachnoid hemorrhage in patients aged over 18 years is determined and correlated with clinical course and neurological outcome after 6 month as determined by modified Rankin score. Additionally, patients are monitored for incidence of delayed cerebral ischemia (DCI) and the incidence of new infarction on the discharge ct scan attributable to DCI. General treatment of cerebral aneurysm and subarachnoid hemorrhage in all patients follows international guidelines.

ELIGIBILITY:
Inclusion Criteria:

* confirmed aneurysmal subarachnoid hemorrhage
* admission within 72hours after hemorrhage
* Age >18 years

Exclusion Criteria:

* non-aneurysmal SAH
* admission >72hours after hemorrhage
* Age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with confirmed aneurysmal subarachnoid hemorrhage admitted within 72 hours to our department aged over 18 years.
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2012-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
modified Rankin score | 6 month after discharge

SECONDARY OUTCOMES:
Incidence of DCI related new infarction on discharge ct scan | at discharge, approx. 14-21days after admission
  Incidence of new infarction on discharge ct scan not attributable to causes other then DCI.

CONTACTS AND LOCATIONS:
Overall Officials: Kerim Beseoglu, M.D., Principal Investigator — Department of Neurosurgery, Heinrich-Heine-University, Düsseldorf
Locations (1):
- Department of Neurosurgery, Heinrich-Heine-University Düsseldorf, Düsseldorf, North Rhine-Westphalia, Germany